CLINICAL TRIAL: NCT01001195
Title: Safety and Efficacy of Three Formulations of AGN-210669 Ophthalmic Solution Compared With Bimatoprost Ophthalmic Solution
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 210669-010
Record Dates: First submitted 2009-10-22; First posted 2009-10-26 (Estimated); Results first posted 2013-10-18 (Estimated); Last update posted 2013-10-18 (Estimated); Status verified 2013-08

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Bimatoprost

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- AGN-210669 ophthalmic solution, 0.1% (Experimental): One drop of AGN-210669 ophthalmic solution, 0.1% in both eyes each evening from Day 1 through the evening prior to Day 29. Selected sites: One additional drop in both eyes on Day 29.
  Interventions: Drug: AGN-210669 ophthalmic solution, 0.1%
- AGN-210669 ophthalmic solution, 0.075% (Experimental): One drop of AGN-210669 ophthalmic solution, 0.075% in both eyes each evening from Day 1 through the evening prior to Day 29. Selected sites: One additional drop in both eyes on Day 29.
  Interventions: Drug: AGN-210669 ophthalmic solution, 0.075%
- AGN-210669 ophthalmic solution, 0.05% (Experimental): One drop of AGN-210669 ophthalmic solution, 0.05% in both eyes each evening from Day 1 through the evening prior to Day 29. Selected sites: One additional drop in both eyes on Day 29.
  Interventions: Drug: AGN-210669 ophthalmic solution, 0.05%
- bimatoprost ophthalmic solution 0.03% (Active Comparator): One drop of bimatoprost ophthalmic solution 0.03% in both eyes each evening from Day 1 through the evening prior to Day 29. Selected sites: One additional drop in both eyes on Day 29.
  Interventions: Drug: bimatoprost ophthalmic solution 0.03%

INTERVENTIONS:
Drug: AGN-210669 ophthalmic solution, 0.1% — One drop of AGN-210669 ophthalmic solution, 0.1% in both eyes each evening from Day 1 through the evening prior to Day 29. Selected sites: One additional drop in both eyes on Day 29.
  Arms: AGN-210669 ophthalmic solution, 0.1%
Drug: AGN-210669 ophthalmic solution, 0.075% — One drop of AGN-210669 ophthalmic solution, 0.075% in both eyes each evening from Day 1 through the evening prior to Day 29. Selected sites: One additional drop in both eyes on Day 29.
  Arms: AGN-210669 ophthalmic solution, 0.075%
Drug: AGN-210669 ophthalmic solution, 0.05% — One drop of AGN-210669 ophthalmic solution, 0.05% in both eyes each evening from Day 1 through the evening prior to Day 29. Selected sites: One additional drop in both eyes on Day 29.
  Arms: AGN-210669 ophthalmic solution, 0.05%
Drug: bimatoprost ophthalmic solution 0.03% — One drop of bimatoprost ophthalmic solution 0.03% in both eyes each evening from Day 1 through the evening prior to Day 29. Selected sites: One additional drop in both eyes on Day 29.
  Other Names: LUMIGAN®
  Arms: bimatoprost ophthalmic solution 0.03%

SUMMARY:
This study will evaluate the safety, efficacy and dose-response of AGN-210669. This study will also compare AGN-210669 with bimatoprost ophthalmic solution (LUMIGAN®).

ELIGIBILITY:
Inclusion Criteria:

* Ocular hypertension or primary open-angle glaucoma in each eye
* Patient requires IOP lowering medication in each eye

Exclusion Criteria:

* Ocular hyperemia or other ocular surface findings in either eye
* Active ocular disease
* Current or anticipated use of any topical ocular medication (including artificial tears) during the study
* Intraocular surgery within past six months or unilateral cataract surgery.
* Functionally significant visual field loss
* Anticipated wearing of contact lenses during study
* Use of other medications that affect IOP such as glaucoma treating medications, within 2 months of screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2009-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AGN-210669 Ophthalmic Solution, 0.1% | AGN-210669 Ophthalmic Solution, 0.075% | AGN-210669 Ophthalmic Solution, 0.05% | Bimatoprost Ophthalmic Solution 0.03%
Started | 39 | 41 | 44 | 41
Completed | 37 | 39 | 44 | 41
Not Completed | 2 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AGN-210669 Ophthalmic Solution, 0.1% | AGN-210669 Ophthalmic Solution, 0.075% | AGN-210669 Ophthalmic Solution, 0.05% | Bimatoprost Ophthalmic Solution 0.03% | Total
Number analyzed (Participants) | 39 | 41 | 44 | 41 | 165
Age, Customized [Number; unit: Participants]
  <45 years | 1 | 1 | 2 | 0 | 4
  45 to 65 years | 22 | 24 | 21 | 21 | 88
  >65 years | 16 | 16 | 21 | 20 | 73
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 22 | 23 | 18 | 87
  Male | 15 | 19 | 21 | 23 | 78

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Eye Intraocular Pressure (IOP)
Description: IOP is a measurement of the fluid pressure inside the eye. The average of the 2 eyes is used for the analyses. A negative number change from baseline indicates a reduction in IOP (improvement) and a positive number change from baseline indicates an increase in IOP (worsening).
Time Frame: Baseline, Day 29 Hour 0
Population: Modified Intent to Treat: all randomized and treated patients who had at least a baseline visit and 1 postbaseline IOP evaluation
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | AGN-210669 Ophthalmic Solution, 0.1% | AGN-210669 Ophthalmic Solution, 0.075% | AGN-210669 Ophthalmic Solution, 0.05% | Bimatoprost Ophthalmic Solution 0.03%
Number analyzed (Participants) | 39 | 41 | 44 | 41
Millimeters of Mercury (mmHg)
  Baseline - Hour 0 | 25.88 (3.696) | 25.18 (2.382) | 25.39 (2.770) | 25.73 (3.490)
  Change from Baseline at Day 29 - Hour 0 | -7.50 (4.219) | -7.65 (3.171) | -5.66 (3.082) | -8.57 (3.854)

ADVERSE EVENTS:
Description: The Safety Population consisted of all randomized and treated patients and was used to assess adverse events (AEs) and serious adverse events (SAEs).
Arm/Group | AGN-210669 Ophthalmic Solution, 0.1% | AGN-210669 Ophthalmic Solution, 0.075% | AGN-210669 Ophthalmic Solution, 0.05% | Bimatoprost Ophthalmic Solution 0.03%
Serious Adverse Events (participants affected / at risk) | 1/39 | 0/41 | 0/44 | 0/41
Other Adverse Events (participants affected / at risk) | 28/39 | 35/41 | 23/44 | 29/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AGN-210669 Ophthalmic Solution, 0.1% (N=39) | AGN-210669 Ophthalmic Solution, 0.075% (N=41) | AGN-210669 Ophthalmic Solution, 0.05% (N=44) | Bimatoprost Ophthalmic Solution 0.03% (N=41)
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AGN-210669 Ophthalmic Solution, 0.1% (N=39) | AGN-210669 Ophthalmic Solution, 0.075% (N=41) | AGN-210669 Ophthalmic Solution, 0.05% (N=44) | Bimatoprost Ophthalmic Solution 0.03% (N=41)
Conjunctival Hyperaemia (Eye disorders) | 21 | 23 | 13 | 25
Punctate Keratitis (Eye disorders) | 5 | 3 | 4 | 3
Photophobia (Eye disorders) | 4 | 5 | 2 | 1
Eye Pain (Eye disorders) | 3 | 4 | 0 | 1
Vision Blurred (Eye disorders) | 2 | 5 | 2 | 1
Foreign Body Sensation in Eyes (Eye disorders) | 2 | 4 | 0 | 1
Anterior Chamber Cell (Eye disorders) | 2 | 1 | 1 | 0
Eye Irritation (Eye disorders) | 2 | 1 | 0 | 2
Instillation Site Pain (General disorders) | 2 | 1 | 0 | 1
Eye Pruritus (Eye disorders) | 0 | 1 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.